CLINICAL TRIAL: NCT04954638
Title: The Effectiveness of Hyperpure Chlorine Dioxide and Sodium Hypochlorite Irrigants During Endodontic Retreament on the Healing of Chronic Periapical Lesions - Clinical, Radiological and Microbiological Study. Randomized Clinical Trial.
Brief Title: The Effectiveness of Hyperpure Chlorine Dioxide and Sodium Hypochlorite Irrigants in Endodontic Retreament in RCT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Eniko Vaszine Szabo (Other)
Responsible Party: Sponsor-Investigator, Eniko Vaszine Szabo, principal investigator, Semmelweis University
Organization: Semmelweis University (Other)
Other Study IDs: OGYÉI/39205/2018
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Persistent Infection; Periapical Lesion
Keywords: hyperpure chlorine dioxide; sodium hypochlorite
MeSH Terms: conditions — Persistent Infection | interventions — Sodium Hypochlorite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen Description microbiological samples taken during the mechanical removal of the root canal obturation using paper points and endodontic files without human DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sodium hypochlorite: group 1: control group with sodium hypochlorite desinfection
  Interventions: Other: endodontic desinfection
- hyperpure chlorine dioxide: group 2: study group with hyperpure chlorine dioxide desinfection
  Interventions: Other: endodontic desinfection

INTERVENTIONS:
Other: endodontic desinfection — * outcome assessment of the retreatment of endodontically treated teeth presenting chronic apical periodontitis
  * effectiveness of hyperpure chlorine dioxide compared with sodium hypochloride
  * using microbiological methods
  * outcome assessed by radiological method and clinical evaluation
  Other Names: hyperpure chlorine dioxide, sodium hypochlorite

SUMMARY:
Endodontic treatment aims to eliminate pathogenic microbes from the root canal. Hyperpure chlorine dioxide is an endodontic irrigant. Our goal is to compare the efficacy of hyperpure chlorine dioxide with the gold standard sodium hypochlorite in the non-surgical retreatment of root canal treated teeth with chronic periapical lesions in a randomized clinical trial. Forty patients having chronic apical periodontitis will randomly be chosen for the study from the patients attending our Department of Conservative Dentistry. Endodontic treatment will be done according to professional quidelines. The patients will randomly be divided into two groups. In the first (control) group sodium hypochlorite, in the second group hyperpure chlorine dioxide will be used as desinfectant. The first sample will be taken from the root canal after removing the previous root canal obturation prior to desinfection. The second sample will be taken one week after temporization. The samples will be evaluated by culturing, MALDI-ToF and PCR strip test. After root canal obturation the the periapical status will be followed by clinical evaluation and control x-rays.

DETAILED DESCRIPTION:
Endodontic treatment aims to eliminate pathogenic microbes from the root canal. This is an almost impossible task as microbes, especially Enterococci are able to line the dentin tubules that are nearly unaccessable to desifectants used during treatment. Hyperpure chlorine dioxide is an endodontic irrigant. In vitro studies proved it to be a very potent desinfectant against which bacteria do not produce resistency. It selectively binds to three amino acids targeting bacterial cells. Due to its small molecular weight and its highly volatile characteristics we presume that it is able to penetrate into the small dentin tubuli. There have been many in vitro studies comparing its characteristics and efficacy, but there have been no in vivo studies done to approve its clinical preformance so far. Our goal is to compare the efficacy of hyperpure chlorine dioxide with the gold standard sodium hypochlorite in the non-surgical retreatment of root canal treated teeth with chronic periapical lesions in a randomized clinical trial. Its efficacy will be compared by microbiological methods and by clinical and radiological evaluation. According to our hypothesis hyperpure chlorine dioxide is more effective antimicrobial agent than the gold standard sodium hypochlorite. The protocol for this clinical study was approved by the Hungarian National Ethics Committee for clinical trials. Forty patients having chronic apical periodontitis will randomly be chosen for the study from the patients attending our Department of Conservative Dentistry. Written consent will be collected from the patients. Only those patients will be accepted who had the root canal treatment done more than four years ago, the tooth is asymptomatic, functionally and esthetically restorable, the coronal restoration can be done within 3-4 weeks of the root canal obturation, who will not have prosthetic or orthodontic treatment interfering with the radiological follow-up and have no general medical conditions or medication influencing the healing of the periapical lesion. Endodontic treatment will be done according to professional quidelines. After sterilizing the tooth and its environment, a sterility test will be be done by taking samples from the top of the restoration (S1) and from the pulp chamber (S2). The root canal obturation will be removed mechanically and a microbiological sample will be taken from the root canal (M1). After taking the sample from the root canal the tooth will be chemomechanically prepared. The patients will randomly be divided into two groups. In the first (control) group sodium hypochlorite, in the second group hyperpure chlorine dioxide will be used as desinfectant. The sample taking procedure will be repeated after one week of temporization (sterility tests S3, S4 and root canal sample M2). The samples will be cultured and identified by MALDI-ToF MS. The remaining samples will be used for PCR testing (Micro-IDent Plus11, Hain Lifescience) to determine the presence of the tested bacteria. In the second session the root canal obturation will be completed. Following coronal restoration a control x-ray will be done by using an individual bite-block for standardization. The success of the root canal treatment will be followed-up by evaluating the periapical status with the Periapical Index scoring system and clinical evaluation according to the criteria set by the European Society of Endodontology including pain assessment where the patients rate pain on the VNRS, with 0 = ''no pain'' to 10 = ''worst pain imaginable". Clinical evaluation and control x-rays will be done at 6 months, 1, 2, 3, and 4 years following treatment. The x-rays will be evaluated by two blinded calibrated examiners.

ELIGIBILITY:
Inclusion Criteria:

• patients having asymptomatic chronic apical periodontitis of size 4-5 according to periapical index scoring system

Exclusion Criteria:

* patients who suffer from diabetes, osteoporosis, cancer, autoimmue disease
* patients who are in immune suppressed state
* patients receiving steroid, bisphosphonate, denosumab or antiangiogenic therapy
* alcoholism
* smoking
* patients having had antibiotic therapy in the past 4 weeks before starting treatment
* teeth with furcation involvement
* teeth with deeper than 4 mm probing depth or the same on neighboring teeth
* patients intending to undergo prosthodontic or orthodontic treatment within four years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients attending the clinic
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Microbiological assessment | 4 years
  The presence of bacteria will be assessed in microbiological samples will be taken from the root canal prior to root canal desinfection after removing obturation and one week after desinfection before obturation. They will be quantified by culturing and specified by MALDI ToF MS. The same samples will be used for PCR strip test to spcify certain test bacteria.
Radiological assessment | 4 years
  After coronal restoration is completed a control x-ray will be taken by means of an individual bite-block. The periapical status will be assessed at the time of obturation-restoration, 6 months, 1, 2, 3, 4 years following endodontic treatment. The outcome will be determined according to the Periapical Index scoring system. The teeth will be evaluated according to healed, healing or unsuccessful as outcome.
Clinical evaluation | 4 years
  At each control appointments a clinical evaluation will be done according to the criteria set by the European Society of Endodontology including: presence of fistula and/or swelling, functionality.
Clinical evaluation | 4 years
  pain evaluated by visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Enikő Vasziné Szabó, DMD PhD, Principal Investigator — Semmelweis University; Zsolt Lohinai, DMD PhD, Study Director — Semmelweis University
Locations (1):
- Semmelweis University, Dental Faculty, Conservative Dentistry Department, Budapest, Hungary